CLINICAL TRIAL: NCT02970526
Title: Evaluation of Intensity and Consequences of Neuropathic Disorders Induced by Oxaliplatin in Patients After Chemotherapy: Observational and Cross-sectional Study
Brief Title: Long Term Effect of Oxaliplatin Treatment in Cancer Survivors
Acronym: PREVOX
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0290
Record Dates: First submitted 2016-11-18; First posted 2016-11-22 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2019-01

CONDITIONS: Colorectal Cancer Survivors; Oxaliplatin Regimen; Adult
Keywords: Colorectal cancer survivors
MeSH Terms: interventions — Oxaliplatin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- colorectal cancer survivors
  Interventions: Drug: Oxaliplatin

INTERVENTIONS:
Drug: Oxaliplatin — Intensity of neuropathy induced by oxaliplatin evaluated by the QLQ-CIPN20 Questionnaire (EORTC).

SUMMARY:
This project will evaluate the neurotoxic effects of oxaliplatin. Oxaliplatin is considered the most neurotoxic chemotherapy, and at the origin of peripheral neuropathies. These neuropathies remain a problem in oncology because currently no prevention strategy has proved effective and only duloxetine seems to have a therapeutic benefit in improving symptoms. In the case of oxaliplatin, neuropathy forced oncologists to reduce the dose or to stop the chemotherapy, potentially degrading the oncological prognosis.

Objective of this study will be to assess, on a large number of patients (n> 500) who completed adjuvant chemotherapy (FOLFOX), the intensity of neuropathic disorders out of 5 years after the end of chemotherapy. Furthermore, this study should enable an assessment of the relationship between the intensity of neuropathy and comorbidities, such as anxiety and depression and health related quality of life of patients.

DETAILED DESCRIPTION:
Oxaliplatin remains the reference treatment of advanced colorectal cancer and more broadly of digestive cancers, incorporated in the FOLFOX protocol (folinic acid, 5-Fu, Oxaliplatin). But oxaliplatin chemotherapy is certainly the most neurotoxic, as on average 90% of patients develop acute neuropathic disorders (within hours or days of the infusion) and 30% to 50% of patients develop a chronic neuropathy with repeated cycles of chemotherapy. The neuropathic grade and duration of symptoms remain variable across studies. Although symptoms improve with time, long-term studies suggest a persistent neuropathy beyond 24 months. Moreover, Vatandoust and colleagues suggest that chemotherapy-induced neuropathy is more frequent and severe over the long term (≥ 12 months) than in previous works published.

In cancer survivors, neuropathy induced by oxaliplatin has a deleterious impact on their quality of life. But, few studies are available on the consequences of oxaliplatin-induced neuropathy in these patients, while these patients remain, in 2003, the third largest group of cancer survivors.

Only 7 studies have specifically evaluated neuropathic disorders induced by oxaliplatin after chemotherapy. Moreover, as pointed Vatandoust and colleagues, there is a real need to understand the long term effects of this chemotherapy-induced neuropathy. More specifically, only two studies have evaluated the effects of neuropathy on quality of life and comorbidities of patients.

Objective of this study will be to assess, on a large number of patients (n> 500) who completed adjuvant chemotherapy (FOLFOX), the intensity of neuropathic disorders out of 5 years after the end of chemotherapy. Furthermore, this study should enable an assessment of the relationship between the intensity of neuropathy and comorbidities, such as anxiety and depression and health related quality of life of patients.

ELIGIBILITY:
Inclusion Criteria:

* • Living patient who received adjuvant chemotherapy (FOLFOX).

  * Patient in remission.
  * FOLFOX chemotherapy over for 0-5 years.
  * Oral Non-opposition to participation in the study

Exclusion Criteria:

* • Patient unable to understand or respond to questionnaires.

  * Age <18 years.
  * Neurological diseases (eg Parkinson's disease, stroke, fibromyalgia ...).
  * Legal incapacity (person deprived of liberty or under guardianship).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: colorectal cancer survivors
Sampling Method: Non-Probability Sample
Enrollment: 409 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

PRIMARY OUTCOMES:
Intensity of neuropathy induced by oxaliplatin evaluated by the QLQ-CIPN20 Questionnaire (EORTC). | once and until 5 years after the end of chemotherapy

SECONDARY OUTCOMES:
Thermal hypersensitivity to cold and hot assessed by VAS. | once and until 5 years after the end of chemotherapy
Neuropathic pain evaluated by the DN4 interview questionnaire. | once and until 5 years after the end of chemotherapy
Anxiety and depression assessed by HADS questionnaire. | once and until 5 years after the end of chemotherapy
Health related quality of life assessed by QLQ-C30 questionnaire (EORTC). | once and until 5 years after the end of chemotherapy
Grade of neuropathy during chemotherapy (NCI-CTCAE). | once and until 5 years after the end of chemotherapy
Cumulative dose (mg / m²) and dose intensity (mg / m² / week) of oxaliplatin | once and until 5 years after the end of chemotherapy
pain assessed by visual analog scale (VAS). | once and until 5 years after the end of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Denis PEZET, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Background] Selvy M, Pereira B, Kerckhove N, Gonneau C, Feydel G, Petorin C, Vimal-Baguet A, Melnikov S, Kullab S, Hebbar M, Bouche O, Slimano F, Bourgeois V, Lebrun-Ly V, Thuillier F, Mazard T, Tavan D, Benmammar KE, Monange B, Ramdani M, Pere-Verge D, Huet-Penz F, Bedjaoui A, Genty F, Leyronnas C, Busserolles J, Trevis S, Pinon V, Pezet D, Balayssac D. Long-Term Prevalence of Sensory Chemotherapy-Induced Peripheral Neuropathy for 5 Years after Adjuvant FOLFOX Chemotherapy to Treat Colorectal Cancer: A Multicenter Cross-Sectional Study. J Clin Med. 2020 Jul 27;9(8):2400. doi: 10.3390/jcm9082400. PMID 32727095
- [Derived] Balayssac D, Kerckhove N, Selvy M, Pereira B, Gonneau C, Petorin C, Vimal-Baguet A, Melnikov S, Kullab S, Hebbar M, Bouche O, Slimano F, Bourgeois V, Lebrun-Ly V, Thuillier F, Mazard T, Tavan D, Benmammar KE, Monange B, Ramdani M, Pere-Verge D, Huet-Penz F, Bedjaoui A, Genty F, Leyronnas C, Pezet D, Martin V. Motor disorders related to oxaliplatin-induced peripheral neuropathy: long-term severity and impact on quality of life. Support Care Cancer. 2024 Jun 13;32(7):427. doi: 10.1007/s00520-024-08627-8. PMID 38869647